CLINICAL TRIAL: NCT03347994
Title: A Phase I Pilot Study of Minnelide, A Novel Heat Shock Protein 70 Inhibitor, in Adult Patients With Relapsed or Refractory Acute Myeloid Leukemia
Brief Title: Minnelide in Adult Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Discordance in contractual language and terms.
Sponsor: Justin Watts (Other)
Collaborators: Minneamrita Therapeutics LLC (Industry)
Responsible Party: Sponsor-Investigator, Justin Watts, Assistant Professor of Medicine, University of Miami
Organization: University of Miami (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170643
Record Dates: First submitted 2017-11-15; First posted 2017-11-20 (Actual); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Acute Myeloid Leukemia
Keywords: Acute Myeloid Leukemia; AML; Refractory AML; Relapsed AML; Refractory Acute Myeloid Leukemia; Relapsed Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — 14-O-phosphonooxymethyltriptolide disodium salt; Injections

STUDY DESIGN:
Intervention Model Description: Dose escalation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Minnelide 0.40 (Dose Level -1) (Experimental): Dose Level -1: 25% decrease from prior dose level
  - 0.40 mg/m2 administered intravenously on days 1-5, 8-12, and 15-19 of a 28 day cycle
  Interventions: Drug: Minnelide
- Minnelide 0.53 (Dose Level 1) (Experimental): Starting Dose Level 1:
  * 0.53 mg/m2 administered intravenously on days 1-5, 8-12, and 15-19 of a 28 day cycle
  Interventions: Drug: Minnelide
- Minnelide 0.67 (Dose Level 2) (Experimental): Dose Level 2: 25% increase from Dose Level 1
  - 0.67 mg/m2 administered intravenously on days 1-5, 8-12, and 15-19 of a 28 day cycle
  Interventions: Drug: Minnelide
- Minnelide 0.80 (Dose Level 3) (Experimental): Dose Level 3: 25% increase from Dose Level 2
  - 0.80 mg/m2 administered intravenously on days 1-5, 8-12, and 15-19 of a 28 day cycle
  Interventions: Drug: Minnelide

INTERVENTIONS:
Drug: Minnelide — Minnelide therapy may be administered for up to 12 cycles of 28 days are planned. If patients are receiving clinical benefit, treatment can continue beyond 12 cycles.
  Other Names: Minnelide for Injection

SUMMARY:
Minnelide, a water-soluble disodium salt variant of triptolide, is a diterpenoid heat shock protein 70 (HSP70) inhibitor. Studies using AML cell lines, primary patient samples, and mouse transplant models demonstrate that Minnelide has potent cell killing effects. Minnelide has already been developed for human use and given to patients in a phase I trial for gastrointestinal (GI) cancers. Given the clinical safety profile and preliminary activity described in human GI cancers, the low-nanomolar anti-leukemic potency of triptolide in vitro, and that minnelide doses predicted to be significantly below the maximum tolerated dose (MTD) in human GI cancers decreased leukemia burden in animal models, the investigators propose a phase I trial in acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is a Phase 1, open label, dose-escalation, safety, pharmacokinetic, and pharmacodynamic pilot study of minnelide given to adult patients with relapsed or refractory AML.

The patient population will consist of adults previously diagnosed with relapsed/refractory AML for whom standard curative or life-prolonging treatment is unavailable or is no longer effective. Patients who are on hydroxyurea may be included in the study and may continue on hydroxyurea while participating in this study.

Once enrolled into the study, patients will be administered Minnelide via a 30-minute IV infusion. Each 28-day treatment cycle is composed of 5 consecutive daily doses of Minnelide followed by a 2-day rest period, repeating for 21 days, followed by a 7-day rest period.

Minnelide therapy may be administered for up to at least 12 cycles provided that the patient tolerates treatment and there is evidence of clinical benefit. If patients are still receiving clinical benefit, treatment may continue beyond 12 cycles, depending on drug availability and drug manufacturer (Minneamrita®) agreement. Study drug may be discontinued early if a patient experiences study drug related toxicities. Patients may discontinue therapy at any time. Patients will attend an End-of-Study visit 30 (+/- 10) days after receiving their last dose of study drug.

To determine the MTD of minnelide, an approach using traditional "3+3" escalation rules will be used. Dose-limiting toxicity (DLT) will be defined as events that are considered by the investigator to be related to therapy with minnelide. Although DLTs may occur at any point during treatment, only DLTs occurring during Cycle 1 of treatment will influence decisions regarding dose escalation. The initial minnelide dose will be 0.53 mg/m2 per dose; (3 dose levels will be explored; 0.53 mg/m2, 0.67 mg/m2, and 0.80 mg/m2). If more than 1 DLT occurs at Dose Level 1, then the next dose to be evaluated (Dose Level -1) will be 0.40 mg/m2. If more than 1 DLT occurs at Dose Level -1, the investigators will consider stopping the study. More conservative dose escalation, evaluation of intermediate doses, and expansion of an existing dose level are all permissible at the discretion of the investigator, if such measures are needed for patient safety or for a better understanding of the dose-related toxicity, exposure, or pharmacodynamics of minnelide.

Toxicity will be evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.0. Adverse events (AEs) will be assessed, and laboratory values, vital signs, and electrocardiograms (ECGs) will be obtained to evaluate the safety and tolerability of minnelide. Serial blood samples for determination of the plasma concentration of minnelide will be obtained during Cycle 1 at pre-specified time points. Assessment of disease response will follow the criteria outlined in the recommendations of the International Working Group (IWG) for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in myeloid malignancies [21, 22]. Circulating leukemic blasts will be assayed for pharmacodynamic marker levels before and at pre-defined time points after minnelide administration to characterize the extent and duration of the biological effects of minnelide in leukemic cells. Exploratory analyses of potential relationships between measures of plasma drug exposure and pharmacodynamic effects of minnelide may be performed as permitted by the data.

ELIGIBILITY:
Inclusion Criteria:

1. Relapsed or refractory Acute Myeloid Leukemia (AML) as defined by International Working Group (IWG) criteria. (Therapy-related AML and/or secondary AML evolving from an antecedent hematologic disorder are not excluded).
2. Adult patients 18 years of age or older
3. Ability to understand the investigational nature, potential risks and benefits of the research study and to provide valid written informed consent.
4. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
5. Patients must satisfy the following laboratory criteria:

   1. Total bilirubin ≤ 1.5 x upper limit of normal (ULN) except in patients with Gilbert's syndrome. Patients with Gilbert's syndrome may enroll if direct bilirubin is ≤ 2 x upper limit of normal of direct bilirubin.
   2. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) must be ≤ 2.5 × ULN
   3. Creatinine 1.5 x ULN or calculated creatinine clearance > 50ml/min
   4. White blood cell (WBC) count < 50,000/µL before administration of Minnelide on Cycle 1 Day 1. Note: Hydroxyurea may be used to suppress the WBC to < 50,000/µL to qualify patients for the study, during the study hydroxyurea may be used for the first 28 days of treatment according to the investigator's discretion.
6. Suitable venous access to allow for all study related blood sampling (safety and research)
7. Estimated life expectancy, in the judgment of the Investigator, which will permit receipt of at least six weeks of treatment
8. Able to understand and willing to sign written informed consent and HIPAA documents
9. Female patients who are postmenopausal for at least one year before the screening visit OR surgically sterile OR of childbearing potential.
10. Agree to practice one highly effective method and one additional effective (barrier) method of contraception, at the same time, from the time of signing the informed consent through 4 months after the last dose of study drug (female and male condoms should not be used together), OR agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.
11. Male patients, even if surgically sterilized (i.e., status postvasectomy), who agree to practice effective barrier contraception during the entire study treatment period and through four months after the last dose of study drug (female and male condoms should not be used together), OR agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence [e.g., calendar, ovulation, symptothermal, postovulation methods for the female partner], withdrawal, spermicides only, and lactational amenorrhea are not acceptable methods of contraception.
12. Able to undergo bone marrow aspiration or biopsy at screening

Exclusion Criteria:

1. Therapy with any investigational products, systemic anti-neoplastic therapy, or radiotherapy within 14 days prior to Cycle 1 Day 1. Patients actively receiving hydroxyurea are eligible and may continue to receive hydroxyurea during protocol treatment.
2. Candidates for standard and/or potentially curative treatments. (A candidate is defined as a patient that is both eligible and willing to have these treatments.)
3. Major surgery within 28 days prior to Cycle 1 Day 1
4. New York Heart Association Class III or IV heart failure, myocardial infarction within the past 6 months, unstable arrhythmia, or evidence of ischemia on ECG
5. Baseline corrected QT interval (QTc) exceeding 480 msec using the Fridericia formula and/or patients receiving class 1A or class III antiarrythmic agents.
6. Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
7. Known, active HIV, Hepatitis A, B or C infection (prior Hepatitis C infection that has been treated and determined to be cured is allowed)
8. Female patients who are pregnant or breast feeding. (Confirmation that the patient is not pregnant will require a negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test result obtained during screening; pregnancy testing is not required for post-menopausal or surgically sterilized women.)
9. Females of child bearing potential who refuse to either practice two effective methods of contraception at the same time or abstain from heterosexual intercourse from the time of signing the informed consent through four months after the last dose of study drug
10. Males of child bearing potential who either refuse to practice effective barrier contraception or abstain from heterosexual intercourse during the entire study treatment period and through four months after the last dose of study drug. (Includes surgically sterilized males - i.e., status post vasectomy)
11. Female patients who are both lactating and breastfeeding, or have a positive serum pregnancy test during the screening period or a positive urine pregnancy test on Day 1 before first dose of study drug
12. Female patients who intend to donate eggs (ova) during the course of this study or within four months after receiving their last dose of study drug(s)
13. Male patients who intend to donate sperm during the course of this study or within four months after receiving their last dose of study drug(s)
14. Significant medical or psychiatric disorder likely in the judgment of the Investigator to interfere with compliance to protocol treatment/research
15. Symptomatic central nervous system (CNS) involvement with leukemia
16. A concurrent second active and non-stable malignancy. Patients with a concurrent second active but stable malignancy are eligible.
17. Known hepatic cirrhosis or severe pre-existing hepatic impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-04 (Estimated); Primary Completion 2021-04 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Safety Profile of Minnelide: Rate of Toxicity in Study Participants | From first dose of therapy to within 30 days after final dose; assessed up to 13 months
  Rate of toxicity in study participants including serious adverse events (SAEs), grade 3 or higher adverse events (AEs), and dose limiting toxicities (DLTs) by treatment dose level cohorts. Toxicity will be assessed in terms of nature, grade and attribution to treatment, using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE), Version 4.03.
  * Evaluable for Safety: Study participants who receive at least one dose of Minnelide therapy.
  * Evaluable for DLT: Study participants who either experience a DLT during Cycle 1 or receive at least 12 (80%) of scheduled doses of minnelide during Cycle 1 without a DLT. Missed doses will not be made up. Eligible patients who discontinue minnelide therapy, miss more than 3 doses of Minnelide, or require a dose reduction in minnelide during Cycle 1 for reasons other than DLT will not be evaluable for DLT and will be replaced.
Maximum Tolerate Dose (MTD) of Minnelide | During Cycle 1, up to 28 days
  The MTD will be defined as highest dose level below or at the maximally administered dose for which ≤ 1 out of 6 patients experiences a dose-limiting toxicity (DLT). To determine the MTD of Minnelide, an approach using traditional "3+3" escalation rules will be used. Dose-limiting toxicity (DLT) will be defined as events that are considered by the investigator to be related to therapy with minnelide. Although DLTs may occur at any point during treatment, only DLTs occurring during Cycle 1 of treatment will influence decisions regarding dose escalation.
Recommended Phase 2 Dose (RP2D) of Minnelide | During Cycle 1, up to 28 days
  Following the proposed dose escalation and expansion cohort, the RP2D of Minnelide will be established as the highest dose level tested for which no more than 2 out of 12 patients experiences a dose-limiting toxicity.

SECONDARY OUTCOMES:
Efficacy of Minnelide Therapy: Overall Response Rate (ORR) | Disease assessment at Baseline, Cycle 2 Day 1, afterwards on Day 1 of each/every other 28-day cycle at investigator discretion, End of Study; Assessed up to 13 months
  Efficacy will be determined by overall response rate (ORR) to Minnelide therapy in study participants. Overall response rate includes rate of study participants experiencing complete response (CR), CR with incomplete bone marrow recovery (CRi); or Partial response (PR) to Minnelide therapy. Best response will be determined using serial blood and bone marrow sampling throughout the course of treatment. Responses will be documented according to revised/modified International Working Group (IWG) Response Criteria (Cheson et al. 2003 for AML and update 2010). Study participants who receive at least 1 cycle of protocol therapy, have measurable disease at baseline, and have at least one post-baseline disease assessment are evaluable for efficacy.
Pharmacokinetics (PK): Area Under the Curve (AUC) of Plasma Concentration of Minnelide | Cycle 1 Days 1, 2, 8 and 9
  The area under the plasma concentration-time curve from time 0 to 24 hours post-dose (AUC24hr) will be assessed. Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize Cmax for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacokinetics (PK): Maximum (Peak) Plasma Concentration (Cmax) of Minnelide | Cycle 1 Days 1, 2, 8 and 9
  Cmax is the maximum (or peak) plasma concentration that a drug achieves in a specified compartment or test area of the body after the drug has been administrated and before the administration of a second dose. Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize Cmax for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacokinetics (PK): Time to maximum plasma concentration (Tmax) of Minnelide | Cycle 1 Days 1, 2, 8 and 9
  Tmax is the time it takes a drug or other substance to reach the maximum concentration (Cmax). Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize Tmax for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacokinetics (PK): Terminal Phase Half Life (t1/2) of Plasma Concentration of Minnelide | Cycle 1 Days 1, 2, 8 and 9
  Terminal phase half-life (t1/2) will be assessed. Half-life (t1/2) is the amount of time it takes for the drug concentration in the plasma to decline by half. Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize terminal phase half life for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacokinetics (PK): total body clearance (CL/F) | Cycle 1 Days 1, 2, 8 and 9
  Apparent total clearance of the drug from plasma, the rate at which a drug is removed from the body, considered as a single unit, the sum of renal clearance + hepatic clearance + other clearance, expressed as volume per unit time. Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize terminal phase half life for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacokinetics (PK): Apparent Volume of Distribution (Vd/F) | Cycle 1 Days 1, 2, 8 and 9
  The apparent volume of distribution is the theoretical volume of fluid into which the total drug administered would have to be diluted to produce the concentration in plasma. Serial blood samples for the determination of plasma concentrations of Minnelide will be collected at pre-specified time points during Cycle 1 to characterize the PK of Minnelide. Plasma for measuring Minnelide concentrations will be collected on day 1 and 8 pre-dose, at the end of infusion (EOI), 0.5, 2, 4, 6, 24 hours post-dose. Descriptive statistics will be used to summarize terminal phase half life for each dose level and all patients. Study participants who receive at least 1 dose of minnelide therapy and undergo at least 5 PK blood draws with concentration-time data to reliably estimate PK parameters are evaluable for PK.
Pharmacodynamics (PD): Expression and Activity Levels of HSP70, PI3K/Akt/mTOR, MAPK/ERK pathway and other relevant markers | Assessed up to 12 months
  Pharmacodynamic (PD) measurements will be obtained from serial blood and bone marrow sampling at specified time points to describe the PD effects of Minnelide. PD paramaters include HSP70 expression and activity, mitochondrial cytochrome c, caspase-3 activation, PI3K/Akt/mTOR and MAPK/ERK pathway activity, and other relevant markers. Study participants who receive at least 1 dose of Minnelide and undergo at least 2 PD blood and bone marrow samples are evaluable. Descriptive statistics will be used to summarize PD parameters for each dose level and all patients.
  * Blood - PD Sampling at pre-dose Cycle 1 Day 1, Day 2 and Day 8; at investigator discretion afterwards on Day 1 of each/every other cycle , and End of Study visit; assessed up to 12 months
  * Marrow - PD Sampling at pre-dose Cycle 1 Day 1, Cycle 2 Day 1; at investigator discretion afterwards and End of Study visit; assessed up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Justin Watts, MD, Principal Investigator — University of Miami